CLINICAL TRIAL: NCT04370665
Title: A Pilot Study for Brain Delivery of Cerezyme® in Patients With Parkinson's Disease Using MR-guided Focused Ultrasound Induced Opening of the Blood-brain Barrier
Brief Title: Blood-Brain-Barrier Disruption With Cerezyme in Patient's With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PD013
Record Dates: First submitted 2020-04-15; First posted 2020-05-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
Keywords: Exablate; Focused Ultrasound
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm, open-labelled study to enroll six (6) patients with Parkinson's disease for three biweekly deliveries of Cerezyme® to the unilateral putamen corresponding to the most affected side using Exablate and Definity®-induced BBB opening. This is a dose escalation study. Each subject will be followed for three months after the final procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label single arm (Experimental): Using Exablate Model 4000 Type-2 to temporarily disrupt the blood brain barrier to deliver Cerezyme in patients with Parkinson's Disease.
  Interventions: Device: Exablate BBBD with Cerezyme

INTERVENTIONS:
Device: Exablate BBBD with Cerezyme — Blood Brain Barrier Disruption via Exablate to deliver Cerezyme.
  Other Names:
  Exablate Neuro

SUMMARY:
This clinical trial focus on the delivery of Cerezyme® in Parkinson's Disease (PD) patients using MR-guided focused ultrasound (MRgFUS) induced opening of the blood-brain barrier (BBB).

DETAILED DESCRIPTION:
Leveraging the preclinical evidence and clinical experience with MRgFUS BBB opening in human subjects, the investigators propose a phase I open-label study to determine the safety and feasibility of three biweekly delivery of Cerezyme® (an analogue of the human enzyme beta-glucocerebrosidase) via MRgFUS induced BBB opening to unilateral putamen in PD. The putamen contains terminals of dopaminergic neurons from the substantia nigra, and is a critically affected brain region in PD. The primary objective is to determine the feasibility of repeated MRgFUS BBB opening for Cerezyme delivery in unilateral putamen. The secondary objective is to describe the safety and tolerability of the procedure. Another objective is to measure changes in PD relevant clinical scores and Cerezyme relevant biomarkers in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between age 35 and 75 years, inclusive.
2. Able and willing to give informed consent.
3. Diagnosis of Parkinson's Disease.
4. At least 2 years from initial diagnosis
5. On stable regiment of PD medications for at least 90 days prior to the study
6. Able to communicate during the Exablate MRgFUS procedure.
7. Able to attend all study visits.

Exclusion Criteria:

1. Previous neurosurgical procedure for PD
2. Cerezyme hypersensitivity
3. Patients who had recent intracranial hemorrhage or stroke
4. Skull covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp. Patients who have clips or other metallic implanted objects in the skull or the brain.
5. Patients who are on blood thinners within washout period prior to treatment (i.e., antiplatelet or vitamin K inhibitor anticoagulants within 7 days, non-vitamin K inhibitor anticoagulants within 72 hours, or heparin-derived compounds within 48 hours of treatment).
6. Patients with a history of a bleeding disorder, blood clotting, coagulopathy or with a history of spontaneous tumor hemorrhage.
7. Patients receiving bevacizumab (Avastin) therapy.
8. Currently participating in another clinical therapeutic trial
9. Documented myocardial infarction within six months of enrollment.
10. Unstable angina on medication.
11. Congestive heart failure.
12. Unstable cardiac arrhythmia.
13. Cardiac pacemaker.
14. Severe hypertension (diastolic BP > 100 on medication).
15. Documented cerebral infarction within the past 12 months or TIA in the past 1 month.
16. Insulin-dependent diabetes mellitus that is not well-controlled or that in the Investigator's opinion precludes participation in the study.
17. Known sensitivity to gadolinium
18. Known sensitivity to DEFINITY ultrasound contrast agent or perflutren.
19. Contraindications to MRI such as non-MRI-compatible implanted devices.
20. Large subjects not fitting comfortably into the MRI scanner.
21. Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia.
22. Untreated, uncontrolled sleep apnea.
23. Positive pregnancy test (for pre-menopausal women).
24. Known life-threatening systemic disease.
25. Severely impaired renal function and/or on dialysis.
26. Right to left or bi-directional cardiac shunt.
27. Subjects with evidence of cranial or systemic infection.
28. Subjects with uncontrolled chronic pulmonary disorders.
29. Subjects with a history of severe asthma, hay fever, or multiple allergies that is not well-controlled (e.g. with anaphylaxis).
30. Subjects with a family or personal history of cardiac arrhythmia.
31. Severe liver injury.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement on MR imaging | Immediately after MRgFUS BBBD procedure
  MRgFUS BBB Opening will be determined qualitatively by contrast enhancement in the sonicated putamen on T1-weighted with gadolinium MRI, and quantitatively by the change in intensity relative to contralateral unsonicated putamen immediately after MRgFUS BBBD procedure.

SECONDARY OUTCOMES:
Safety --Adverse events | Through study completion, an average of 3 months
  Safety will be assessed by recording all adverse events and/or Serious Adverse Events that are BBBD related. Each Adverse Event will be documented for patterns of occurrence.

OTHER OUTCOMES:
Exploratory effectiveness of Cerezyme delivery via MRgFUS BBB Opening | 1 day after the final BBBD procedure
  Exploratory effectiveness of Cerezyme delivery via MRgFUS BBB Opening will be measured by changes in levels of Cerezyme (GCase) and GCase substrates levels (e.g. GL1 and glucosylsphingosine or lyso-GL1) in cerebralspinal fluid (CSF) samples.
Exploratory effectiveness of Cerezyme treatment via MRgFUS BBB Opening | 3 months after the final BBBD procedure.
  Exploratory effectiveness of Cerezyme treatment via MRgFUS BBB Opening will be measured by changes in cognitive impairment via Mini-Mental Status Exam (MMSE).

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada